CLINICAL TRIAL: NCT01375322
Title: Efficacy and Safety of Two Fixed-combination Antihypertensive Regimens, Amtrel® and Co-Diovan® in Type 2 Diabetes Hypertension Patients With Microalbuminuria
Brief Title: ADDM Study - Amtrel and Co-Diovan in Type 2 Diabetes Mellitus Hypertension Patients With Microalbuminuria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TSH Biopharm Corporation Limited (Industry)
Responsible Party: Owen Chen/Clinical Research Manager, TSH Biopharm Corporation Limited
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTY-ABM-0601
Record Dates: First submitted 2011-06-15; First posted 2011-06-17 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Hypertension; Diabetes Mellitus, Type 2; Albuminuria
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Albuminuria | interventions — benazepril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Co-Diovan® Group (Active Comparator): The starting dose of Co-Diovan® was 1 capsule (contains 1/2 tablet) (valsartan/ hydrochlorothiazide 40 mg/ 6.25 mg) every morning and could be adjusted up to 2 capsules (contains 1 tablet per capsule) (valsartan/ hydrochlorothiazide 160 mg/ 25.0 mg) every morning if patients did not achieve the criteria of SBP<130 mmHg and DBP< 80 mmHg during treatment period
  Interventions: Drug: Valsartan+Hydrochlorothiazide
- Amtrel® Group (Experimental): The starting dose of Amtrel® was 1 capsule (contains 1/2 tablet) (amlodipine / benazepril hydrochloride 2.5 mg/ 5 mg) every morning and could be adjusted up to 2 capsules (contains 1 tablet per capsule) (amlodipine / benazepril hydrochloride 10 mg/ 20 mg) every morning if patients did not achieve the criteria of SBP<130 mmHg and DBP< 80 mmHg during treatment period
  Interventions: Drug: Amlodipine+Benazepril

INTERVENTIONS:
Drug: Amlodipine+Benazepril — Amlodipine besylate 5 mg + Benazepril hydrochloride 10 mg, daily use and forced titrate till 16-week end
  Other Names: Amtrel®
  Arms: Amtrel® Group
Drug: Valsartan+Hydrochlorothiazide — Valsartan 80 mg + Hydrochlorothiazide 12.5 mg, daily use and forced titrate till 16-week end
  Other Names: Co-Diovan®
  Arms: Co-Diovan® Group

SUMMARY:
The purpose of the study is to compare the change from baseline in blood pressures (DBP/SBP) to 16-week regimen between Amtrel® and Co-Diovan®. The secondary objectives were listed as the following.

* To compare the response rate (defined as SBP < 130 mmHg and DBP < 80 mmHg) at the end of study
* To evaluate the change from baseline in albumin-to-creatinine ratio with antihypertensive medications in whole group (combined treatment groups) and each treatment group (Amtrel®, Co-Diovan®) at Week 16
* The change from baseline in glycosylated hemoglobin (HbA1c) at Week 16
* The change from baseline in fasting plasma glucose (FPG) at Week 16
* The change from baseline in fasting lipid profiles (triglyceride, total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol) at Week 16
* The change from baseline in arteriosclerosis marker (brachial-ankle pulse-wave velocity (ba-PWV) and ankle-brachial pressure index (ABI), using Colin-VP1000) at Week 16
* The change from baseline on the body mass index (BMI) and waist-hip ratio (WHR) at each specified study time point
* To ascertain the safety and tolerability of Amtrel® versus Co-Diovan® including AE/SAE, and laboratory examinations

DETAILED DESCRIPTION:
At the screening visit, patients who fulfilled the entrance criteria and had given written informed consent entered a placebo running period where they discontinued antihypertensive medication for two weeks. During that period, Adalat 5mg could be given for emergency. At the end of placebo running period those patients became hypertensive (i.e., SBP between 130-180mmHg or DBP between 80-110mmHg) were randomized into either treatment group. For those patients remaining normotensive continued to be on placebo run-in for another two weeks (10 - 14 days). After the two-week (10 - 14 days) placebo run-in period those patients became hypertensive were randomized into either treatment group. However for those patients remaining normotensive were excluded from the study. After randomization into either arm, patients entered four months treatment period. The dosage adjustment were proceed in order to reach the best effect. During the treatment period there was a monthly visit to assess the response of the patients.

The starting dose of Amtrel® was 1 capsule (contains 1/2 tablet) (amlodipine / benazepril hydrochloride 2.5 mg/ 5 mg) every morning and could be adjusted up to 2 capsules (contains 1 tablet per capsule) (amlodipine / benazepril hydrochloride 10 mg/ 20 mg) every morning if patients did not achieve the criteria of SBP<130 mmHg and DBP< 80 mmHg during treatment period.

The starting dose of Co-Diovan® was 1 capsule (contains 1/2 tablet) (valsartan/ hydrochlorothiazide 40 mg/ 6.25 mg) every morning and could be adjusted up to 2 capsules (contains 1 tablet per capsule) (valsartan/ hydrochlorothiazide 160 mg/ 25.0 mg) every morning if patients did not achieve the criteria of SBP<130 mmHg and DBP< 80 mmHg during treatment period.

All randomized patients attended monthly clinic visits for the 16-week treatment period. At week 4 (Visit 3), all patients were force-titrated to 1 capsule (1 tablet per capsule) for 4 weeks. Subsequently, those patients did not achieve the target blood pressure (SBP<130 mmHg and DBP<80 mmHg) were titrated monthly to next dose level (2 capsule per day).

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes with stable controlled (HbA1c between 6.5-10%)
* SBP between 130-180mmHg or DBP between 80-110mmHg
* microalbuminuria (UAE 30-300mg/24hrs or creatinine 30-300mg/g)

Exclusion Criteria:

* IDDM or secondary forms of diabetes
* hepatic and/or renal dysfunction
* serum potassium level > 5.5mmol/L
* severe renal disease
* Chronic Heart Failure (NYHA class III or IV)
* unstable CV disease
* PTCA within 3 months

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2007-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To compare the change from baseline in blood pressures (DBP/SBP) to 16-week regimen between Amtrel® and Co-Diovan® | 16-week

SECONDARY OUTCOMES:
To compare the response rate (defined as SBP < 130 mmHg and DBP < 80 mmHg) at the end of study | 16-week

CONTACTS AND LOCATIONS:
Overall Officials: Wayne H-H Sheu, Principal Investigator — Taichung Veterans General Hospital
Locations (4):
- Taiwan (4):
  - Chang Gung Memorial Hospital-Kaohsiung, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Tri-Service General Hospital, Taipei
  - Far Eastern Memorial Hospital, Taipei

REFERENCES:
- [Derived] Lee IT, Hung YJ, Chen JF, Wang CY, Lee WJ, Sheu WH. Comparison of the efficacy and safety profiles of two fixed-dose combinations of antihypertensive agents, amlodipine/benazepril versus valsartan/hydrochlorothiazide, in patients with type 2 diabetes mellitus and hypertension: a 16-week, multicenter, randomized, double-blind, noninferiority study. Clin Ther. 2012 Aug;34(8):1735-50. doi: 10.1016/j.clinthera.2012.06.014. Epub 2012 Jul 10. PMID 22784975